CLINICAL TRIAL: NCT01619748
Title: Effects of Obstructive Sleep Apnoea and Its Treatment on Macrovascular and Microvascular Function
Brief Title: Peripheral Vascular Function in Obstructive Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: STH-16309
Record Dates: First submitted 2012-06-08; First posted 2012-06-14 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Obstructive Sleep Apnoea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Untreated OSA patients: Patients with obstructive sleep apnoea who are untreated
- OSA patients highly compliant with CPAP: OSA patients established on CPAP therapy (high compliance, > 80% nightly use for ≥ 4 h per night)
- OSA patients poorly compliant with CPAP: OSA patients established on CPAP therapy (poor compliance, 10% < nightly use < 50% or < 4 h per night)
- Age and BMI-matched controls: Age and BMI-matched controls without OSA

SUMMARY:
Peripheral vascular function is impaired in people with obstructive sleep apnoea who are untreated compared with age-, weight- and sex-matched healthy controls.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a chronic respiratory disorder associated with endothelial dysfunction, increased sympathetic activation and increased cardiovascular risk. The standard treatment paradigm is continuous positive airway pressure (CPAP), however, patient adherence to CPAP is variable. It is unclear to what extent that poor adherence to CPAP therapy augments vascular endothelial function and reduces cardiovascular risk compared to excellent adherence. The main aim of this research is to investigate vascular endothelial function in OSA patients who are poorly-adherent to CPAP therapy. Nitric oxide (NO)-mediated, endothelium-dependent macrovascular and microvascular function (by brachial artery flow-mediated dilatation and forearm cutaneous thermal hyperaemia, respectively) and generalised microvascular function (by post-occlusion reactive hyperaemia) will be assessed in three obese OSA patient populations (high-adherence (n=20); low adherence (n=20); and, untreated (n=20)) and age-/BMI-matched OSA-free controls. We will also assess body composition, cardiovascular risk, lipid status and functional capacity. This research will evaluate treatment efficacy in patients who are poorly-adherent to CPAP treatment and could identify whether an alternative approach to their care should be explored.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnoea diagnosed using overnight polysomnography
* Age 18-90 years

Exclusion Criteria:

* Unable to perform the tests involved in the study
* Unable to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and controls living in and around Sheffield, UK
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation of the brachial artery | Baseline only
  The brachial artery dilator response to a 5-min period of forearm arterial occlusion will be measured using a vascular ultrasound scanner and a 7-MHz linear array probe.

SECONDARY OUTCOMES:
GTN-mediated dilatation of the brachial artery | Baseline only
  The brachial artery vasodilator response to a 400 microgram sublingual dose of glyceryl trinitrate will be measured using vascular ultrasound imaging.
Forearm skin blood flow response to 5-min proximal-cuff arterial occlusion | Baseline only
  Proximal arterial occlusion will be performed by inflating a blood pressure cuff placed on the upper arm to 200 mmHg for 5 min. After cuff deflation, the skin blood flow response will be measured using laser Doppler flowmetry.
Forearm skin blood flow response to localised heating at 42 degrees C | Baseline only
  A local heating unit on the forearm will be heated from 33 to 42 degrees C at a rate of 1 degree C every 10 s. Temperature will be held at 42 degrees C for 35 min. The increase in skin blood flow will be measured using a laser Doppler flowmetry probe placed in the centre of the local heating unit.

CONTACTS AND LOCATIONS:
Overall Officials: Garry A Tew, PhD, Study Director — Sheffield Hallam University; James Moss, BSc, Principal Investigator — Sheffield Hallam University; Stephen Bianchi, MD, Study Director — Sheffield Teaching Hospitals NHS FT
Locations (2):
- United Kingdom (2):
  - Centre for Sport and Exercise Science, Sheffield Hallam University, Sheffield, South Yorkshire
  - Sheffield Teaching Hospitals NHS FT, Sheffield, South Yorkshire